CLINICAL TRIAL: NCT01475370
Title: Study of OCV-501 in Patients With Acute Myeloid Leukemia (AML) (Extension From Study 311-10-001)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 311-10-002; JapicCTI-111646 (Other: JAPIC)
Record Dates: First submitted 2011-10-18; First posted 2011-11-21 (Estimated); Results first posted 2021-03-02 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute myeloid leukemia; WT1
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OCV-501 (Experimental)
  Interventions: Drug: OCV-501

INTERVENTIONS:
Drug: OCV-501 — 1. Before the recommended dose will be decided OCV-501 will be subcutaneously administered once a week at the dose in the study 311-10-001.
  2. After the recommended dose will be decided OCV-501 will be subcutaneously administered once a week at the recommended dose.

SUMMARY:
The purpose of this study is to assess the safety of OCV-501 in patients with AML who completed the Study 311-10-001 and were judged that there was no relapse by any inspections in the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients who completed the Study 311-10-001 and were judged that there was no relapse by any inspections in the end of the study.
* Patients who are capable of giving informed consent

Exclusion Criteria:

* Patients failed to discontinue the Study 311-10-001 even though patients met the discontinuation criteria.
* Patients who have participated in any other clinical trials , excluding the Study 311-10-001).

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-01-24 (Actual); Primary Completion 2016-12-22 (Actual); Study Completion 2016-12-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center, Tokyo, Japan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was an extension trial from the preceding Trial 311-10-001. Subjects who had undergone the observations, examinations, and evaluations which were stipulated for Trial 311-10-001 and who met all the inclusion criteria and did not fall under any of the exclusion criteria for this trial were selected for this trial.
Groups:
- OCV-501 0.3mg: OCV-501 was subcutaneously administered once a week, with each subject receiving the same dose as in Trial 311-10-001 (i.e. continued administration of 0.3 mg).
- OCV-501 1 mg: OCV-501 was subcutaneously administered once a week, with each subject receiving the same dose as in Trial 311-10-001 (i.e. continued administration of 1 mg).
- OCV-501 3 mg: OCV-501 was subcutaneously administered once a week, with each subject receiving the same dose as in Trial 311-10-001 (i.e. continued administration of 3 mg).
Period: Overall Study
Arm/Group | OCV-501 0.3mg | OCV-501 1 mg | OCV-501 3 mg
Started | 3 | 3 | 3
Completed | 0 | 0 | 0
Not Completed | 3 | 3 | 3
Not completed — Exacerbation of primary disease | 2 | 2 | 2
Not completed — Study drug administration difficult | 0 | 1 | 1
Not completed — Other than specified | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The demographics and other baseline characteristics of subjects enrolled in this trial were the same as those in Trial 311-10-001 as the trial was an extension trial from the preceding Trial 311-10-001 and the data obtained before the start of investigational medicinal product (IMP) administration in Trial 311-10-001 were used as the baseline data in this trial.
Groups:
- Total: Total of all reporting groups
Arm/Group | OCV-501 0.3mg | OCV-501 1 mg | OCV-501 3 mg | Total
Number analyzed (Participants) | 3 | 3 | 3 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1 | 2
  >=65 years | 2 | 3 | 2 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 0 | 4
  Male | 1 | 1 | 3 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 3 | 3 | 3 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 3 | 3 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Relapse of Acute Myeloid Leukemia Based on the International Working Group Response Criteria
Description: Bone marrow samples were taken by bone marrow aspiration, and the percentage of bone marrow blasts was calculated. The result was assessed according to the International Working Group Response Evaluation Criteria where a case was designated as relapse if any of the following occurred: reappearance of leukemic blasts in the peripheral blood or ≥ 5% blasts in the bone marrow after complete response (morphologic relapse).
Time Frame: Treatment period (from the first IMP administration until the time of discontinuation)
Measure: Number; unit: participants
Arm/Group | OCV-501 0.3mg | OCV-501 1 mg | OCV-501 3 mg
Number analyzed (Participants) | 3 | 3 | 3
participants | 2 | 2 | 2

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were collected from the first IMP administration until the time of discontinuation.
Arm/Group | OCV-501 0.3mg | OCV-501 1 mg | OCV-501 3 mg
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 3/3 | 2/3 | 3/3
Other Adverse Events (participants affected / at risk) | 2/3 | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OCV-501 0.3mg (N=3) | OCV-501 1 mg (N=3) | OCV-501 3 mg (N=3)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Acute myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OCV-501 0.3mg (N=3) | OCV-501 1 mg (N=3) | OCV-501 3 mg (N=3)
Ichthyosis (Congenital, familial and genetic disorders) | 0 | 0 | 1
Ear pruritus (Ear and labyrinth disorders) | 1 | 1 | 0
Vertigo positional (Ear and labyrinth disorders) | 1 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 1 | 0 | 0
Dry eye (Eye disorders) | 0 | 1 | 0
Glaucoma (Eye disorders) | 0 | 1 | 0
Hypermetropia (Eye disorders) | 0 | 1 | 0
Dental caries (Gastrointestinal disorders) | 1 | 0 | 1
Injection site reaction (General disorders) | 2 | 2 | 3
Injection site induration (General disorders) | 1 | 2 | 0
Injection site erythema (General disorders) | 0 | 2 | 0
Injection site discolouration (General disorders) | 1 | 1 | 0
Administration site reaction (General disorders) | 1 | 0 | 0
Injection site anaesthesia (General disorders) | 1 | 0 | 0
Injection site mass (General disorders) | 1 | 0 | 0
Injection site pain (General disorders) | 0 | 1 | 0
Injection site pruritus (General disorders) | 0 | 1 | 0
Injection site swelling (General disorders) | 0 | 1 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1
Abscess (Infections and infestations) | 0 | 0 | 1
Cystitis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1
Localised infection (Infections and infestations) | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 1 | 2
White blood cell count decreased (Investigations) | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Post herpetic neuralgia (Nervous system disorders) | 0 | 0 | 1
Sciatica (Nervous system disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Eczema nummular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No